CLINICAL TRIAL: NCT00893711
Title: Lactobacillus Reuteri Versus Placebo in the Treatment and Prevention of Infantile Colic: a Clinical and Microbiological, Double-blind, Prospective, Randomised, Controlled Study
Brief Title: Lactobacillus Reuteri Versus Placebo in the Treatment and Prevention of Infantile Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Dr. SAVINO Francesco, MD, PhD, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FS-2009
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Infantile Colic
Keywords: infantile colic; lactobacillus; gut microflora; FISH; toll like receptor; T reg; messenger RNA; CC-chemokine receptor 7; interleukin 10
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lactobacillus reuteri (Active Comparator): Lactobacillus reuteri DSM 17938 is administered at a dose of 1.000.000.000 colony forming units (CFU) in V drops of a commercially available oil suspension, 30 min before feeding, once a day for 30 days.
  Interventions: Other: Lactobacillus reuteri DSM 17938
- Placebo (Placebo Comparator): Placebo is administered in V drops once a day for 30 days. Placebo is inactive, similar to the studied treatment with the same package, taste, characteristics of colour and consistency.
  Interventions: Other: Placebo
- L.reuteri + vit D (Active Comparator): L. reuteri DSM 17938 (10^8 CFU) plus vitamin D3 (400 UI) five drops/day for 3 months
  Interventions: Dietary Supplement: L.reuteri + Vit D
- Vit D Placebo (Placebo Comparator): vitamin D3 (400 UI) five drops/day for 3 months
  Interventions: Dietary Supplement: Vit D placebo

INTERVENTIONS:
Other: Lactobacillus reuteri DSM 17938 — Lactobacillus reuteri is administered at a dose of 1.000.000.000 colony forming units (CFU) in V drops/day for 21 days
  Other Names: Reuterin,Noos - Italy; BIOGAIA drops - Sweden
  Arms: Lactobacillus reuteri
Other: Placebo — Placebo is administered in V drops once a day for 21 days. Placebo is inactive, similar to the studied treatment with the same package, taste, characteristics of colour and consistency.
  Other Names: Placebo BIOGAIA Sweden
  Arms: Placebo
Dietary Supplement: L.reuteri + Vit D
  Other Names: Reuterin D3 drops, Noos Italy; Reuflor D3 drops, Recordati Italy
  Arms: L.reuteri + vit D
Dietary Supplement: Vit D placebo
  Arms: Vit D Placebo

SUMMARY:
The purpose of this study is:

* to study the intestinal microflora of colicky infants before and after L. reuteri or placebo administration, evaluating the effect of Lactobacillus reuteri on the growth of the main intestinal microbiota (coliforms, Clostridium butyricum, Lactobacilli, Bifidobacteria) with fluorescent in situ hybridization (FISH) technique or with Real-Time PCR Taqman; Further, the global intestinal microflora composition, using large-scale DNA sequencing of 16S rRNA genes ( 454-pyrosequencing technique.
* to evaluate the improvement of colicky symptoms by the oral administration of Lactobacillus reuteri (primary outcome: reduction of the daily average crying time from baseline to the end of the treatment period, to less than 3 hours a day, the cut-off proposed by Wessel; secondary outcome: number of responders versus non-responders in each group at the end of the treatment).
* to evaluate fecal calprotectin values at the beginning and at the end of the study. BÜHLMANN Quantum Blue® Calprotectin High Range (Schönenbuch, Switzerland). A quantitative immunoassay.
* to evaluate Th17/Treg balance at time 0 and t 30 ( days) investigating mRNA FOXP3 and RORγ in peripheral blood using RT-PCR Real Time Taqman.
* the measurement of the expression level of CC-chemokine receptor 7 messenger RNA using the real-time TaqMan reverse transcription polymerase chain reaction method.
* the measurement of expression of interleukin 10 (IL-10) messenger RNA using the real-time TaqMan reverse transcription polymerase chain reaction method.
* Parental satisfaction at the end of the study period ( 30 day ) with a numerc scale from 1 to 10.

DETAILED DESCRIPTION:
Infantile colic is one of the most common problems within the first three months of life. It consists of a behavioural syndrome characterised by paroxysmal, excessive and inconsolable crying without identifiable cause. Although infantile colic is commonly reported and causes appreciable distress for both parents and paediatricians, despite forty years of research, its aetiology still remains unclear. Recently the role of intestinal microflora has growing importance, and a lower count of intestinal lactobacilli has been observed in colicky infants compared to healthy ones. In a recent study we have observed that Lactobacillus reuteri improved colicky symptoms in breast-fed infants within one week of treatment compared to Simethicone, suggesting that probiotics may play a role in infantile colic (Savino F, Pelle E, Palumeri E, Oggero R, Miniero R.Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics 2007; 119:e124-30). The mechanism involved in such finding is only partially understood and, for this reason, we have planned this new study to evaluate not only the clinical improvement but also the microbiological data.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of infantile colic according to Wessel's criteria
* gestational age between 37 and 42 weeks
* age between 4 and 16 weeks
* birth weight between 2500 and 4000 g
* exclusively breastfed

Exclusion Criteria:

* clinical evidence of chronic illness or gastrointestinal disorders
* administration of probiotics and antibiotics

Ages: 4 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Estimated)
Dates: Start 2008-03; Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the daily average crying time from baseline to the end of the treatment period, to less than 3 hours a day, the cut-off proposed by Wessel and number of responders versus non-responders in each group at the end of the treatment | time 0 - 7 - 21 - 30 days
  diary crying Barr

SECONDARY OUTCOMES:
Responders to treatment | 30 day
  was defined as the number of responders in each group on days 7, 14 , 21 and 30 . Responders (defined in the protocol) were those who experienced a decrease in the daily average crying time of 50% from baseline. Diary Crying Barr.
To analyze intestinal microflora | day 0 and day 30
  The intestinal microflora of the infants will be analyzed the effect of the probiotic on selected intestinal microbiota (Escherichia coli, Clostridium butyricum, Lactobacillus, Bifidobacterium), using fluorescent in situ hybridization (FISH) or using with Real-Time PCR Taqman.
Assay of Th17/Treg balance | time 0- 30 days
  For the analyses of mRNA FOXP3 and RORγ in peripheral blood RT-PCR Real Time Taqman will be used

OTHER OUTCOMES:
Preventive effects of L.reuteri on infantile colic | 5 months
  action on: use of pain relieving agents, switch to infant formula, number of paediatric consultations for infantile colic
Fecal calprotectin values | 0-30 days
  BÜHLMANN Quantum Blue® Calprotectin High Range (Schönenbuch, Switzerland). It is a quantitative determination of fecal calprotectin through a sandwich immunoassay.
Parental satisfacion | day 30
  numeric scale from 1to 10

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Savino, MD, PhD, Principal Investigator — Ospedale Infantile Regina Margherita - Dipartimento di Pediatria.S.S.D. SAPI, Torino
Locations (2):
- Italy (2):
  - Ospedale Infantile Regina Margherita, Torino, TO
  - Ospedale Infantile Regina Margherita, Torino

IPD SHARING:
Plan to Share IPD: Yes
to partecipe to an individual partecipant data meta- analysis.

REFERENCES:
- [Background] Savino F. Focus on infantile colic. Acta Paediatr. 2007 Sep;96(9):1259-64. doi: 10.1111/j.1651-2227.2007.00428.x. PMID 17718777
- [Background] Savino F, Pelle E, Castagno E, Palumeri E, Oggero R. Must infants with colic really be hospitalized? Acta Paediatr. 2007 Jul;96(7):1109; author reply 1110. doi: 10.1111/j.1651-2227.2007.00328.x. Epub 2007 May 10. No abstract available. PMID 17498186
- [Background] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238
- [Background] Savino F, Grassino EC, Guidi C, Oggero R, Silvestro L, Miniero R. Ghrelin and motilin concentration in colicky infants. Acta Paediatr. 2006 Jun;95(6):738-41. doi: 10.1080/08035250500522654. PMID 16754557
- [Background] Savino F, Palumeri E, Castagno E, Cresi F, Dalmasso P, Cavallo F, Oggero R. Reduction of crying episodes owing to infantile colic: A randomized controlled study on the efficacy of a new infant formula. Eur J Clin Nutr. 2006 Nov;60(11):1304-10. doi: 10.1038/sj.ejcn.1602457. Epub 2006 May 31. PMID 16736065
- [Background] Savino F, Castagno E, Bretto R, Brondello C, Palumeri E, Oggero R. A prospective 10-year study on children who had severe infantile colic. Acta Paediatr Suppl. 2005 Oct;94(449):129-32. doi: 10.1111/j.1651-2227.2005.tb02169.x. PMID 16214780
- [Background] Savino F, Cresi F, Castagno E, Silvestro L, Oggero R. A randomized double-blind placebo-controlled trial of a standardized extract of Matricariae recutita, Foeniculum vulgare and Melissa officinalis (ColiMil) in the treatment of breastfed colicky infants. Phytother Res. 2005 Apr;19(4):335-40. doi: 10.1002/ptr.1668. PMID 16041731
- [Background] Savino F, Bailo E, Oggero R, Tullio V, Roana J, Carlone N, Cuffini AM, Silvestro L. Bacterial counts of intestinal Lactobacillus species in infants with colic. Pediatr Allergy Immunol. 2005 Feb;16(1):72-5. doi: 10.1111/j.1399-3038.2005.00207.x. PMID 15693915
- [Background] Savino F, Cresi F, Pautasso S, Palumeri E, Tullio V, Roana J, Silvestro L, Oggero R. Intestinal microflora in breastfed colicky and non-colicky infants. Acta Paediatr. 2004 Jun;93(6):825-9. PMID 15244234
- [Derived] Savino F, Garro M, Montanari P, Galliano I, Bergallo M. Crying Time and RORgamma/FOXP3 Expression in Lactobacillus reuteri DSM17938-Treated Infants with Colic: A Randomized Trial. J Pediatr. 2018 Jan;192:171-177.e1. doi: 10.1016/j.jpeds.2017.08.062. Epub 2017 Sep 29. PMID 28969887
- [Derived] Roos S, Dicksved J, Tarasco V, Locatelli E, Ricceri F, Grandin U, Savino F. 454 pyrosequencing analysis on faecal samples from a randomized DBPC trial of colicky infants treated with Lactobacillus reuteri DSM 17938. PLoS One. 2013;8(2):e56710. doi: 10.1371/journal.pone.0056710. Epub 2013 Feb 28. PMID 23468874